CLINICAL TRIAL: NCT04778176
Title: Assessing the Pharmacokinetics, Safety, Tolerability and Efficacy of Continuous Oral Levodopa Via the DopaFuse® Delivery System in Parkinson's Disease Patients
Acronym: SCOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SynAgile Corporation (Industry)
Collaborators: Clintrex Research Corporation (Unknown); TFS Trial Form Support (Industry); Clinical Data Science GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0007
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DopaFuse Delivery System 50mg LD/hr or 68mg LD/hr flow rate (Experimental): Either 50mg/13mg LD/CD per hour or 68mg/17mg LD/CD per hour flow rate based upon Subject's standard levodopa (LD) dose. Subjects will routinely wear each container for approximately 5 hours (3 containers per day).
  Interventions: Combination Product: continuous oral delivery of levodopa/carbidopa

INTERVENTIONS:
Combination Product: continuous oral delivery of levodopa/carbidopa — The system consists of a reusable custom dental retainer, its case, and a pre-filled, single-use container which continuously releases levodopa/carbidopa into the back of the mouth.

SUMMARY:
The purpose of this study is to evaluate whether the DopaFuse System can reduce the fluctuation of plasma levodopa levels compared to participants' standard intermittent doses of oral LD/CD tablets (background treatment). It will also assess whether the system is safe, well tolerated, and can relieve motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's Disease consistent with UK Brain Bank Criteria
2. Age at least 30 years old at time of consent
3. Male and Female participants (Women of child-bearing potential (WOCB) are eligible for participation if they are not pregnant or breastfeeding and agree to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 30 days after the last dose of study treatment)
4. Suitable for oral retainer wear
5. A good response to Levodopa, as assessed by the Investigator
6. At least 2 hours of wearing OFF time per day, as reported by the participant
7. Predictable early morning OFF periods, in the judgement of the participant and the Investigator
8. Taking 400-1,200 mg of LD/CD per day in at least 4 doses, with stable dosing for the last 28 days prior to screening.
9. A modified Hoehn and Yahr of ≤ 3 in the ON state at screening
10. A stable regimen of anti-PD medications for the last 28 days prior to Screening
11. A Mini-Mental State Examination (MMSE) Score ≥26
12. Capable of giving signed informed consent
13. Approved for entry into the study by the Enrollment Authorization Committee (EAC)

Exclusion Criteria:

1. Atypical or secondary Parkinson's Disease
2. Severe Dyskinesia that might interfere with study performance in the judgement of Investigator
3. Clinically significant dysphagia or sialorrhea that might interfere with administration of study intervention in the judgement of the Investigator
4. Use of extended release levodopa within 28 days prior to screening
5. Any clinically significant medical, surgical, or psychiatric condition; laboratory value or ECG result which, in the opinion of the Investigator, makes the participant unsuitable for study entry or potentially unable to complete all aspects of the study.
6. Presence of clinically significant orthostatic hypotension at screening, in the opinion of Investigator or the EAC
7. Suicidal ideation within 1 year prior to the Screening Visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or attempted suicide within the last 5 years.
8. History of psychosis or hallucinations in the past six months
9. Any malignancy in the past 5 years (excluding basal cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated.)
10. Current or previous diagnosis of malignant melanoma or the presence of any suspicious skin lesion based on physical exam findings
11. Unable to give blood required for the study
12. History of allergic reaction to plastics
13. LD infusion therapy (i.e. Duodopa); current or previous continuous apomorphine infusion treatment.
14. Participation in any other clinical trial <30 days prior to screening visit.
15. Presence of two third molars ("wisdom teeth") on the upper dentition
16. Participants who, for any reason, are judged by the Investigator or the EAC to be inappropriate for this study, including participants who are unable to communicate or cooperate with the Investigator or who have/had a clinically significant illness or abnormal physical examination that may compromise safety of the participant during the trial or affect ability of the participant to adhere to study procedures.
17. Participants taking non-selective monoamine oxidase (MAO) inhibitors
18. Participants with known hypersensitivity to the active ingredients (levodopa, carbidopa) or excipients (Benzoic Acid, Disodium Edetate, Medium Chain Triglycerides, Poloxamer 188) of the drug paste
19. Participants with narrow-angle glaucoma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Variability in plasma concentration of levodopa as assessed with the Levodopa Fluctuation Index (Cmax-Cmin)/Caverage) | pre-dose and every 30 minutes for 12 hours on Days 1 and 2.
  Comparing Day 2 to Day 1 in steady state (4-12 hours). Fluctuation index will also be calculated by the hour.
Treatment Emergent Adverse Events | Screening to Day 29
Serious Adverse Events | Screening to Day 29
Treatment Emergent Adverse Events leading to discontinuation | Screening to Day 29
Percent of participants that complete study | Screening to Day 29
Difference in OFF time between Days 1 and 15, based on in-person investigator ratings | Day 1 compared to Day 15
  Investigator-rated assessment of motor state (ON or OFF) pre-dose and every 30 minutes for 12 hours.

SECONDARY OUTCOMES:
Coefficient of variation (CV) for plasma levodopa. | pre-dose and every 30 minutes for 12 hours on Days 1 and 2.
  This will be calculated between 4 and 12 hours on Days 1 and 2 comparing DopaFuse and oral levodopa tablets.
Variability in plasma concentration of levodopa as assessed with the Levodopa Fluctuation Index (Cmax-Cmin)/Caverage). | pre-dose and every 30 minutes for 12 hours on Days 1 and 2. Pre-dose and at 30 minute intervals for two hours, and at one-hour intervals for the remainder of the 12 hours on Day 3.
  Comparing Day 3 to Day 1, as well as Day 2 (0-12 hours) to Day 1. Fluctuation index will also be calculated by the hour.
Levodopa and Carbidopa peak plasma concentration (Cmax) | pre-dose and every 30 minutes for 12 hours on Days 1 and 2. Pre-dose and at 30 minute intervals for two hours, and at one-hour intervals for the remainder of the 12 hours on Day 3.
Variability in plasma levodopa comparing Dopafuse and oral levodopa tablets based on fluctuation index and CV in participants who are H. pylori negative/positive | pre-dose and every 30 minutes for 12 hours on Days 1 and 2. Pre-dose and at 30 minute intervals for two hours, and at one-hour intervals for the remainder of the 12 hours on Day 3.
Questionnaire for Impulse Control Disorders in Parkinson's Disease Rating Scale (QUIP-RS) | Screening to Day 29
Columbia - Suicide Severity Rating Scale (C-SSRS) | Screening to Day 29
Difference in OFF Time between Day 1 and Day 3 | Day 1 and Day 3
  Investigator-rated assessment of motor state (ON or OFF) pre-dose and every 30 minutes for 12 hours.
Difference in ON Time without troublesome dyskinesia between Days 1, 3 and 15 | Days 1, 3, and 15
  Investigator-rated assessment of motor state (ON or OFF) pre-dose and every 30 minutes for 12 hours.
Difference in ON Time with troublesome (severe) dyskinesia between Days 1, 3 and 15 | Days 1, 3 and 15
  Investigator-rated assessment of motor state (ON or OFF) pre-dose and every 30 minutes for 12 hours.
Change in Unified Parkinson's Disease Rating Scale Part III at 6 hours after morning dose between Days 1, 3 and 15 | Days 1, 3 and 15
Levodopa and Carbidopa time to maximum plasma concentration (Tmax) | pre-dose and every 30 minutes for 12 hours on Days 1 and 2. Pre-dose and at 30 minute intervals for two hours, and at one-hour intervals for the remainder of the 12 hours on Day 3.
Levodopa and Carbidopa area under the plasma concentration versus time curve (AUC) | pre-dose and every 30 minutes for 12 hours on Days 1 and 2. Pre-dose and at 30 minute intervals for two hours, and at one-hour intervals for the remainder of the 12 hours on Day 3.

OTHER OUTCOMES:
A comparison of the subgroups who are H. pylori positive and negative will be performed as an exploratory analysis. | Screening to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim Heller, MBA, Study Chair — SynAgile Corporation
Locations (5):
- Italy (3):
  - San Raffaele Cassino, Cassino
  - Centro Parkinson, Policlinico Tor Vergata, Rome
  - IRCCS San Raffaele Pisana, Rome
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Neuroscience Centre (CINAC), Móstoles, Spain

IPD SHARING:
Plan to Share IPD: No